CLINICAL TRIAL: NCT04421781
Title: Salvage HIFU for Local Recurrence in the Prostatic Bed After Prostatectomy and External Beam Radiation Therapy : Preliminary Results
Acronym: Salvage HIFU
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20_086
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Salvage Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Salvage HIFU for local recurrence after prostatectomy and EBRT: Between July 2005 and November 2018, at Edouard Herriot Hospital (Lyon, France), 22 consecutive patients were treated with S-HIFU for a local recurrence after RP and salvage or adjuvant EBRT. The oncological outcomes (treatment failure-free survival, progression-free survival), the adverse events and urinary incontinence were retrospectively reviewed.
  Interventions: Other: Retrospectively review of medical data in patients treated by Salvage HIFU for isolated macroscopic recurrence in the prostatic bed after radical prostatectomy and salvage or adjuvant EBRT

INTERVENTIONS:
Other: Retrospectively review of medical data in patients treated by Salvage HIFU for isolated macroscopic recurrence in the prostatic bed after radical prostatectomy and salvage or adjuvant EBRT — Patients were treated using dedicated post-EBRT parameters (5-s pulse, 5-s waiting period, 90% of the acoustic power). Between July 2005 and November 2018, at Edouard Herriot Hospital (Lyon, France), 22 consecutive patients were treated with S-HIFU for a local recurrence after RP and salvage or adjuvant EBRT. The oncological outcomes (treatment failure-free survival, progression-free survival), the adverse events and urinary incontinence were retrospectively reviewed.

SUMMARY:
Retrospective monocentric analysis performed on patients treated with salvage HIFU for isolated macroscopic recurrence in the prostatic bed after radical prostatectomy and salvage or adjuvant EBRT. The oncological outcomes (treatment failure-free survival, progression-free survival), the adverse events and urinary incontinence will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patient treated by S-HIFU for a single recurrence within the prostatic bed after an initial RP with curative intent with or without lymphadenectomy followed by salvage or adjuvant EBRT (with or without pelvic lymph node irradiation) combined or not with ADT;

  * life expectancy of ≥10 years;
  * histological local recurrence (positive biopsy),
  * negative metastatic evaluation (All patients underwent multiparametric MRI (mpMRI) to confirm the relapse in the prostatic bed and Choline PET/CT to exclude metastasis (lymph node, visceral or bone metastasis).
  * the use of ADT at BF after S-EBRT was not an exclusion criterion (ADT was introduced by the centre referring the patient).
  * no limits were placed on prostate cancer characteristics, PSA (value, doubling time (PSA-DT)), Gleason score and location of suspected recurrence in relation to the sphincter.

Exclusion Criteria:

* patients who do not meet the inclusion criteria

Ages: 60 Years to 86 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between July 2005 and November 2018, at Edouard Herriot Hospital (Lyon, France), 22 consecutive patients were treated with S-HIFU for a local recurrence after radical prostatectomy and salvage or adjuvant EBRT. The oncological outcomes (treatment failure-free survival, progression-free survival), the adverse events and urinary incontinence were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Oncological outcomes in the prostatic bed after S-HIFU for a local recurrence after RP and salvage or adjuvant EBRT. | December 31, 2019
  Oncological outcomes:
  * Treatment failure-free survival: absence of:
    * recurrent prostate cancer in the prostatic bed and/or
    * metastasis and/or
    * introduction of systemic treatment
  * Progression-free survival: absence of:
    * metastasis and/or
    * introduction of systemic treatment
  * decrease in PSA value: any drop in PSA after S-HIFU, regardless of whether there was subsequent PSA progression
  * BCR-free survival following S-HIFU defined as an absence of two rises in PSA ≥0.2 ng/mL above nadir
  Functional outcomes:
  * complications (Clavien classification)
  * Urinary incontinence (Ingelman-Sundberg score)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology and Transplantation Surgery, Edouard Herriot Hospital,, Lyon, France